CLINICAL TRIAL: NCT02822183
Title: Online Survey of Clinicians to Learn About Their Interpretation of Capnography Waveforms
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Lara Brewer, Research Assistant Professor, University of Utah
Other Study IDs: IRB_00066043
Record Dates: First submitted 2016-06-25; First posted 2016-07-04 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Clinical Interpretation of Capnography Waveforms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Online Survey

SUMMARY:
This online survey presents capnography waveforms and asks the survey participants to give feedback about their interpretation of the patient status, both in the form of a score and a set of text to describe their interpretation.

DETAILED DESCRIPTION:
The capnography waveforms presented were originally collected from patients in various clinical settings, with patients both intubated and non-intubated. The de-identified waveforms are presented along with a statement about whether the patients were intubated or not, the amount of supplemental oxygen provided, and in some cases, the oxygen saturation of hemoglobin in the blood (SpO2). The participants are asked to provide a score between 1 and 10 to indicate their interpretation of the wellbeing of the patient. The participants are also asked to provide up to two sentences of text to describe their interpretation of the patient condition based on the information provided.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians who have at least two years of experience in interpreting capnography waveforms in their clinical practice

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinicians who have at least two years of experience in interpreting capnography waveforms in their clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Wellbeing score | 1 day (survey completion)
Text messages selected by survey participant | 1 day (survey completion)
  Up to two statements describing the interpretation of the condition. For all survey participants, the most commonly preferred text messages will be identified

IPD SHARING:
Plan to Share IPD: No